CLINICAL TRIAL: NCT02731729
Title: A Randomized, Phase 2 Study of Ipilimumab vs Ipilimumab Plus Nivolumab in Patients With Stage III-IV Melanoma Who Have Progressed or Relapsed on PD-1 Inhibitor Therapy
Brief Title: Ipilimumab vs Ipilimumab Plus Nivolumab in Patients With Stage III-IV Melanoma Who Have Progressed or Relapsed on PD-1 Inhibitor Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Parker Institute for Cancer Immunotherapy (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PICI0001; 16-043 (Other: Memorial Sloan Kettering Cancer Center)
Record Dates: First submitted 2016-04-04; First posted 2016-04-07 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Melanoma
Keywords: Ipilimumab; Nivolumab; Stage III-IV Melanoma; Progressed or Relapsed on PD-1 Inhibitor Therapy; 16-043
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Nivolumab

ARMS (2):
- ipilimumab and nivolumab (Experimental): For patients in the combination arm, nivolumab will first be administered intravenously at a dose of 1 mg/kg of body weight over a period of 60 minutes, once every 3 weeks for four doses. Thirty minutes after the completion of each nivolumab infusion, patients will receive 3 mg/kg of ipilimumab over a period of 30 minutes.
  Interventions: Drug: ipilimumab; Drug: nivolumab
- ipilimumab (Experimental): In the ipilimumab monotherapy group, patients will receive 3 mg/kg of ipilimumab over a period of 30 minutes once every 3 weeks for four doses.
  Interventions: Drug: ipilimumab

INTERVENTIONS:
Drug: ipilimumab
  Other Names: Yervoy
Drug: nivolumab
  Other Names: Opdivo
  Arms: ipilimumab and nivolumab

SUMMARY:
The purpose of this research study is to learn whether patients whose disease grows after being treated with nivolumab or pembrolizumab respond to ipilimumab (Yervoy®) alone or in combination with nivolumab (Opdivo®).

ELIGIBILITY:
Main Inclusion Criteria:

1. American Joint Committee on Cancer (AJCC) (2009) Stage IV cutaneous melanoma or Stage III cutaneous, acral or mucosal melanoma that is judged inoperable. Patients with a history of uveal melanoma are not eligible.
2. Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with computerized tomography (CT) scan. Patients must have at least one measurable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) and a separate lesion amenable to biopsy.
3. Histologic proof of melanoma reviewed and confirmed by the enrolling site.
4. Previous treatment with a programmed cell death protein 1 (PD-1) or programmed death-ligand 1 (PD-L1) inhibitor with documented progression of disease on most recent CT scan. Progression of disease is defined as 1) the appearance of a new measureable lesion (>10 mm) on cross-sectional imaging or physical examination OR 2) enlargement of previously detected lesions on two consecutive imaging studies OR 3) enlargement of a previously detected lesion with correlative symptomatology on one cross-sectional imaging study. Patients remain eligible if they had a previous response to a PD-1 inhibitor, including patients who had a complete response, partial response or stable disease (SD). Primary progressing patients are defined as those who received anti-PD-1 therapy within 2 months of study enrollment. Patients with relapsed disease are defined as those who received their last dose of PD-1 blocking antibody ≥2 months prior to enrollment.
5. Patients who received adjuvant PD-1 therapy who then develop measurable disease are eligible. However, they must have received their last dose of PD-1/PD-L1 blockade within two months of enrollment in this study. They will be stratified with patients who have primary progressive disease.
6. Life expectancy of greater than 3 months.
7. Age ≥ 18 years old.
8. Eastern Cooperative Oncology Group performance status = 0 or 1 or Karnofsky Performance Status equivalent.
9. Patients must have adequate organ and marrow function as defined below:

   1. White blood cells >2, 000/microliter (mcL)
   2. Absolute neutrophil count >1,500/mcL
   3. Platelets >100,000/mcL
   4. Hemoglobin > 9.0 g/dL
   5. Total bilirubin ≤ 1.5 X institution's upper limit of normal
   6. Aspartate aminotransferase (serum glutamic oxaloacetic transaminase)/alanine aminotransferase (serum glutamic pyruvic transaminase) ≤ 2.5 X institution's upper limit of normal for patients with no concurrent liver metastases, OR ≤ 5 X institution's upper limit of normal for patients with concurrent liver metastases
   7. Serum creatinine < 1.5x OR creatinine clearance of at least 40
10. Women of childbearing potential must have a negative serum pregnancy test within 24 hours prior to the start of study drug. A woman of childbearing potential is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over age 50 in the absence of other biologic or physiologic causes.
11. Women with child bearing potential and men with reproductive potential must be willing to practice acceptable methods of contraception.
12. Ability to understand and the willingness to sign a written informed consent document.
13. Willingness to undergo biopsy of metastatic site or site of unresectable disease prior to randomization.

Main Exclusion Criteria:

1. History of another malignancy except for those who have been disease-free for 3 years, or patients with a history of completely resected non-melanoma skin cancer and/or patients with indolent secondary malignancies not requiring active therapy, are eligible. Consult the study Medical Monitor if unsure whether second malignancies meet the requirements specified above.
2. Any major surgical procedures or external beam radiotherapy within 14 days prior to study drug administration.
3. Use of other investigational drugs within 28 days prior to study drug administration.
4. Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression. Treated brain metastases must have been stable for at least 1 month and require treatment with less than 10mg/day prednisone equivalent for at least 2 weeks prior to study drug administration.
5. Prior exposure to either ipilimumab or combined checkpoint blockade.
6. Any diagnosis of autoimmune disease. Patients with Type I diabetes mellitus, hypothyroidism only requiring hormone replacement, adrenal insufficiency on replacement dose steroids, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
7. Pregnant women and lactating women.
8. History of uveal melanoma.
9. Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (with the exception of chronic or cleared HBV or HCV infection, which will be allowed). Once-documented negative result for HIV, HBV, and HCV is sufficient.
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection and psychiatric illness/social situations that would limit compliance with study requirements.
11. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted.
12. Patients with history of any grade 4 toxicity during previous anti PD-1 treatment or history of Grade 3 or higher pneumonitis.
13. Patients with a history of Grade ≥2 neuropathy.
14. Prisoners or patients who are involuntarily incarcerated.
15. Children under the age of 18.
16. Patients who require hemodialysis.
17. Patients with a history of allergy to study drug components or history of a severe hypersensitivity reaction to any monoclonal antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2019-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramy Ibrahim, MD, Study Director — Parker Institute for Cancer Immunotherapy
Locations (7):
- United States (7):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Friedman CF, Spencer C, Cabanski CR, Panageas KS, Wells DK, Ribas A, Tawbi H, Tsai K, Postow M, Shoushtari A, Chapman P, Karakunnel J, Bucktrout S, Gherardini P, Hollmann TJ, Chen RO, Callahan M, LaVallee T, Ibrahim R, Wolchok J. Ipilimumab alone or in combination with nivolumab in patients with advanced melanoma who have progressed or relapsed on PD-1 blockade: clinical outcomes and translational biomarker analyses. J Immunother Cancer. 2022 Jan;10(1):e003853. doi: 10.1136/jitc-2021-003853. PMID 35074903
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at four institutions in the United States. Recruitment occurred between June 2016 to May 2018.
Pre-assignment Details: 33 participants were assessed for eligibility. Out of the 33 participants, 20 patients met the inclusion/exclusion criteria and were randomized to the study arms.
Groups:
- Ipilimumab and Nivolumab: For patients in the combination arm, nivolumab will first be administered intravenously at a dose of 1 mg/kg of body weight over a period of 60 minutes, once every 3 weeks for four doses. Thirty minutes after the completion of each nivolumab infusion, patients will receive 3 mg/kg of ipilimumab over a period of 30 minutes.
  ipilimumab
  nivolumab
- Ipilimumab: In the ipilimumab monotherapy group, patients will receive 3 mg/kg of ipilimumab over a period of 30 minutes once every 3 weeks for four doses.
  ipilimumab
Period: Overall Study
Arm/Group | Ipilimumab and Nivolumab | Ipilimumab
Started | 10 | 10
Completed | 1 | 2
Not Completed | 9 | 8
Not completed — Death | 2 | 2
Not completed — Study terminated by Sponsor | 6 | 6
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Out of the 20 patients randomized, one participant randomized to the ipilimumab monotherapy arm withdrew consent before starting treatment. The remaining 19 patients were evaluated for efficacy and safety analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipilimumab and Nivolumab | Ipilimumab | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Median (Full Range); unit: years] | 66 [35 to 83] | 56 [39 to 66] | 60 [35 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 9 | 6 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  White | 7 | 9 | 16
  Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19
ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) Scale of Performance Status is one such measurement. It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). The ECOG Performance Status ranges from 0 (fully active, able to carry on all pre-disease performance without restriction) to 5 (dead).
  Participants
    ECOG Score = 0 | 7 | 6 | 13
    ECOG Score = 1 | 3 | 3 | 6
M stage [Count of Participants; unit: Participants] — The letter "M" indicates whether the cancer has spread to other parts of the body, called distant metastasis. If the cancer has not spread, it is labeled M0. If the cancer has spread, it is considered M1.
  M1a: The cancer has spread to 1 other part of the body beyond the colon or rectum.
  M1b: The cancer has spread to more than 1 part of the body other than the colon or rectum.
  M1c: The cancer has spread to the peritoneal surface.
  Participants
    M0 | 1 | 3 | 4
    M1a | 2 | 1 | 3
    M1b | 3 | 2 | 5
    M1c - without brain metastases | 4 | 3 | 7
Type of Melanoma [Count of Participants; unit: Participants]
  Acral | 1 | 1 | 2
  Cutaneous | 8 | 7 | 15
  Mucosal | 1 | 1 | 2
Genomic Driver [Count of Participants; unit: Participants]
  v-RAF murine sarcoma viral oncogene homolog B1 (BRAF) | 3 | 2 | 5
  Neuroblastoma RAS viral oncogene homolog (NRAS) | 2 | 4 | 6
  Other/Unknown | 5 | 3 | 8
Prior Treatment [Count of Participants; unit: Participants]
  Anti-PD-1 | 10 | 9 | 19
  Other | 3 | 1 | 4
Best response to prior anti-PD-1 treatment [Count of Participants; unit: Participants]
  Stable Disease | 0 | 1 | 1
  Progressive Disease | 9 | 6 | 15
  Unknown | 1 | 2 | 3
Median lactate dehydrogenase [Median (Full Range); unit: units/L] | 214 [157 to 310] | 208 [152 to 1800] | 211 [152 to 1800]
Median time since last anti-PD-1 treatment [Median (Full Range); unit: weeks] | 4.3 [2 to 36] | 6.0 [3 to 55] | 5.1 [2 to 54.7]

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) as Defined by RECIST v1.1 at Week 18
Description: Overall Response Rate was defined as any participant who had a Complete Response (CR) or Partial Response (PR) as defined by RECIST v1.1 by week 18 of treatment.
Time Frame: Week 18
Population: Efficacy-Evaluable Population. The efficacy-evaluable population includes all participants who were randomly allocated to receive either combination ipilimumab/nivolumab or ipilimumab alone and received at least one dose of any study intervention (ipilimumab or nivolumab). For analyses based on this population, participant treatment groups are defined according to the treatment that was assigned at randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipilimumab and Nivolumab | Ipilimumab
Number analyzed (Participants) | 10 | 9
percentage of participants | 20 [3 to 56] | 56 [21 to 86]

2. Secondary Outcome: Disease Control Rate (DCR) Status at Week 18
Description: Disease Control Rate was defined as any participant who achieved a complete response (CR), partial response (PR), or who remained stable (SD) as defined in Recist v1.1 at week 18.
Time Frame: Week 18
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipilimumab and Nivolumab | Ipilimumab
Number analyzed (Participants) | 10 | 9
percentage of participants | 60 [26 to 88] | 67 [30 to 93]

3. Secondary Outcome: Time to Treatment Failure (TTF)
Description: Time to Treatment Failure is defined as the time from treatment initiation until the participant starts a subsequent therapy or death, whichever comes first.
Time Frame: The time from treatment initiation until a subsequent therapy is started or death.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab and Nivolumab | Ipilimumab
Number analyzed (Participants) | 10 | 9
months | 26.9 [0.7 to NA] — The upper confidence limit is not evaluable based on the available data | 13.6 [2.8 to NA] — The upper confidence limit is not evaluable based on the available data

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is defined as the time of treatment initiation to death by any cause
Time Frame: Death
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab and Nivolumab | Ipilimumab
Number analyzed (Participants) | 10 | 9
Participants | 2 | 1

5. Secondary Outcome: Number of Participants With Grade 3 or 4 Adverse Events
Description: The occurrence of Grade 3 and Grade 4 adverse events (AE) assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: AE were monitored during each treatment cycle and could be reported until 30 days after the last dose of study treatment had been administered.
Population: Safety-Evaluable Population. The safety-evaluable population includes all participants who received at least one dose of any study intervention. For analyses based on this population, participant treatment groups will be defined according to the treatment that was assigned at randomization. However, if a participant received the incorrect study drug for the entire period of treatment, the participant's treatment group will be defined as the treatment the participant actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab and Nivolumab | Ipilimumab
Number analyzed (Participants) | 10 | 9
Participants | 4 | 5

6. Secondary Outcome: Disease Control Rate (DCR) Status at Week 12
Description: Disease Control Rate was defined as any participant who achieved a complete response (CR), partial response (PR), or who remained stable (SD) as defined in Recist v1.1 at week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ipilimumab and Nivolumab | Ipilimumab
Number analyzed (Participants) | 10 | 9
Percentage of participants | 60.0 [26.2 to 87.8] | 55.6 [21.2 to 86.3]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during each cycle. Adverse events were reported until 30 days after the last dose of study treatment had been administered.
Arm/Group | Ipilimumab and Nivolumab | Ipilimumab
All-Cause Mortality (participants affected / at risk) | 2/10 | 1/9
Serious Adverse Events (participants affected / at risk) | 2/10 | 4/9
Other Adverse Events (participants affected / at risk) | 10/10 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab and Nivolumab (N=10) | Ipilimumab (N=9)
Colitis (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Reproductive system and breast disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab and Nivolumab (N=10) | Ipilimumab (N=9)
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Hair color changes (Skin and subcutaneous tissue disorders) | 0 | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Nausea (Gastrointestinal disorders) | 5 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 3
Fatigue (General disorders) | 2 | 3
Chills (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 1 | 1
Influenza like illness (General disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 4 | 4
Hypotension (Vascular disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 5 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 1
White blood cell count decreased (Investigations) | 2 | 2
Platelet count decreased (Investigations) | 2 | 1
Weight decreased (Investigations) | 1 | 2
Neutrophil count decreased (Investigations) | 1 | 1
Amylase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Hypophysitis (Endocrine disorders) | 3 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Skin infection (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Proteus infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Vulval disorder (Reproductive system and breast disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Trial Site and/or Co-Principal Investigators may publish or present Study Data and other results of the Study from the Trial Site individually upon the first to occur of: (i) twelve (12) months after conclusion, abandonment, or termination of the Study at all Affiliated Research Institutions, or (ii) after Parker Institute for Cancer Immunotherapy [PICI] confirms in writing there will not be a multi-site Study publication.

DOCUMENTS (2):
  • Study Protocol (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT02731729/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT02731729/SAP_001.pdf